CLINICAL TRIAL: NCT00224978
Title: Chloroquine as Adjuvant to the Treatment of Glioblastoma Multiforme, A Randomized Trial
Brief Title: Chloroquine for Treatment of Glioblastoma Multiforme
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Neurology and Neurosurgery, Mexico (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 14/99
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2009-11-18 (Estimated); Status verified 2009-11

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Chloroquine

INTERVENTIONS:
Drug: Chloroquine

SUMMARY:
Chloroquine is a strong lysosomotropic and DNA-intercalating agent in experimental studies (Neurosurgical Focus 14(2): February, 2003) and an open-label clinical trial the investigators have demonstrated a strong adjuvant effect of chloroquine on the therapy of malignant gliomas. This study will assess in a randomized, placebo-controlled, double-blind study the effects of chloroquine as adjuvant to the conventional therapy of Glioblastoma Multiforme.

DETAILED DESCRIPTION:
ANTECEDENTS: We have shown experimentally a significant adjuvant effect of quinacrine (an analog of chloroquine) on cultured malignant glial cells and C6 implanted malignant glioma in Wistar rats. When quinacrine was added to the standard therapy with carmustine cell destruction and tumor diminution were higher than therapy with carmustine alone. Those results were published in Neurosurgery 2001; 49:969-973 (at that time the manuscript was "in press").

The present protocol started with a controlled, open-label clinical trial on 7 patients with GBM and 7 contemporary control patients. All patients received the same treatment of extensive surgery, carmustine therapy and irradiation at the standard doses as (as described in our previous report Surgical Neurology 2000; 53:157-162). Once selected to enter the study the patients were allocated alternatively in the chloroquine or the control group. Endpoint evaluation was settled as surviving time after the beginning of therapy and the end point follow-up was settled in survivors at two years after the beginning of treatment.

18 months after the beginning of the open trial it was observed that chloroquine treated patients had a longer survival and no adverse effects to chloroquine therapy were seen.

At that time it was decided to start the second part of the protocol designed as a double-blind placebo-controlled trial, ideal number of patients to be included was settled in 15 patients on each group.

The results of the 1st. phase of the study by the open-label trial were published in Neurosurgical Focus (http://www.aans.org/education/journal/neurosurgical/feb03/14-2-3.pdf) on February, 2003.

In order to corroborate the observations (at that time with a short follow-up) of the open trial the double-blind, a placebo-controlled study was initiated in October, 2000; the dose of chloroquine for the blind study was decided to be maintained in 150 mg daily for one year after the beginning of therapy.

The Research Committee was notified on the beginning and the design of this trial: 6,000 tablets of chloroquine 150 mg (Aralen) and 6,000 identical tablets of placebo were commercially purchased and sent to the laboratory of Dr. Roberto Medina at the National Polytechnic Institute (selected as monitor). 30 sets of 375 tablets each were separated (15 contained chloroquine and 15 placebo) in identical flasks, the assignment of treatments was randomly allocated; the codified treatments numbered 1-30 were then sent back to our Institute. The code was sealed and kept by the monitor until the end of the study. Patients included in the study were given the corresponding treatment in sequential order.

Criteria for inclusion of patients in the trial is detailed in methods of the manuscript submitted to the Annals of Internal Medicine Ms. # M0-1087 (pages 6-7).

Follow-up and statistical analysis: End-point evaluation was settled as time of death after the beginning of therapy. Follow-up for survivors was settled at 2 years after the beginning of treatment. Survival distributions were analyzed as a Kaplan-Meier plot and compared by the log rank test. Statistical analysis of demographic, clinical and imaging characteristics of patients was made by the t test for independent values.

After more than four years from the beginning of the study 26 patients from the originally decided goal number of 30 patients had completed at least two years of follow-up. At this time (January 2005) it was decided to open the code and proceed with the analysis of those patients, which turned out to be 13 chloroquine-treated and 13 placebo-treated patients. The last 4 patients (who were not included in the analysis) are currently under treatment but their follow-up will end next year (2 patients are received chloroquine and the other 2 placebo).

No patient initially selected refuse to enter the study, nor any patient included was lost at follow-up. All 26 patients included in the study have been followed until the time of death or up to July 2005 in survivors.

ELIGIBILITY:
Inclusion Criteria:

* Tumor restricted to one hemisphere of the brain
* Karnofsky scale >7
* Histologically confirmed GBM in first or second recurrence or relapse
* Adequate hematologic, hepatic and renal function
* Karnofsky performance status score ≥ 70%
* Life expectancy ≥ 16 weeks

Exclusion Criteria:

* Gastrointestinal dysfunction
* Compromised cardiac function
* Concurrent severe and /or uncontrolled medical conditions

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2005-01; Study Completion 2005-08

PRIMARY OUTCOMES:
Survival after surgery

SECONDARY OUTCOMES:
End-point evaluation, survival at two years

CONTACTS AND LOCATIONS:
Overall Officials: Julio Sotelo, MD, Principal Investigator — National Institute of Neurology and Neurosurgery of Mexico
Locations (1):
- National Institute of Neurology and Neurosurgery, Mexico City, Mexico

REFERENCES:
- [Result] Briceno E, Reyes S, Sotelo J. Therapy of glioblastoma multiforme improved by the antimutagenic chloroquine. Neurosurg Focus. 2003 Feb 15;14(2):e3. doi: 10.3171/foc.2003.14.2.4. PMID 15727424
- [Result] Sotelo J, Briceno E, Lopez-Gonzalez MA. Adding chloroquine to conventional treatment for glioblastoma multiforme: a randomized, double-blind, placebo-controlled trial. Ann Intern Med. 2006 Mar 7;144(5):337-43. doi: 10.7326/0003-4819-144-5-200603070-00008. PMID 16520474